CLINICAL TRIAL: NCT02870166
Title: Genetic Study Explanatory Severe Zinc Deficiencies : Multicenter, Genetics, Controlled and Prospective Study
Brief Title: Genetic Study of Severe Zinc Deficiencies
Acronym: GENEZINC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0193
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Acrodermatitis Enteropathica
MeSH Terms: conditions — Acrodermatitis enteropathica | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sample

SUMMARY:
Given the structural essential, catalytic and co-catalytic played by zinc in many sections of protein metabolism, carbohydrate and lipid (zinc is involved in the function of more than 300 metalloenzymes and metalloproteins), one can imagine the impact of a deficiency or even a sub-chronic zinc deficiency on the health of the individual. Studies multiply that show that, long-term, marginal zinc deficiency is a risk factor for the development of cancer or neurodegenerative complex diseases (eg Alzheimer's disease). In addition, the short-term zinc deficiencies foster the development of skin conditions and susceptibility to viral and bacterial infections. The aim of this project is to identify, in the population of patients with pseudo-acrodermatitis enteropathica (AE) tested in the investigators laboratory, rare variants (mutations "real" epimutations or polymorphisms) located in solute carrier family 39 member 4 (SLC39A4) gene or in 55 other genes chosen for their role in zinc homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Are included all patients (minors included) with suggestive symptoms and biological signs of a hereditary deficiency of zinc, appeared for the first time at birth or weaning (see description given in the introduction);
* Clinical diagnosis of zinc deficiency must be made by a specialist dermatologist, pediatrician or gastroenterologist;
* Zinc deficiency has been audited by an assay of serum zinc, erythrocyte, plasma, urine or hair;
* The response of all symptoms and signs to zinc oral supplementation should be rapid and complete.

Exclusion Criteria:

* All patients with homozygous or compound heterozygous mutations in the SLC39A4 gene are excluded because they have a proven acrodermatitis enteropathica (AE);
* All patients who developed their first symptoms of zinc deficiency outside the neonatal period, most likely because they have an acquired deficiency and not congenital;
* All patients with probable cause of zinc deficiency that is surgery of the digestive tract, chronic digestive disease, or total parenteral nutrition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators had therefore selected 96 individuals for the project. They correspond either to the patients themselves (ie the index case tested in the laboratory) or to mothers and / or fathers of patients who accompany their child consultation. For each of them, the analysis will focus on the genomic DNA was extracted from peripheral blood leukocytes and is stored in the sample bank of DNA laboratory. Note that twenty patients seen by our collaborator neurologist, Prof. Vincent Ramaekers (Belgium) are a subgroup separately in our study, since all have autistic disorders responsive to the zinc, in addition to zinc deficiency. By studying these patients in particular clinical picture, we already approach the possible consequences of zinc deficiency on complex diseases.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Homozygous mutations in the SLC39A4 gene | at 3 years
heterozygous mutations in the SLC39A4 gene | at 3 years
deleterious variants in 55 zinc homeostasis genes in patient | at 3 years
deleterious variants in 55 zinc homeostasis genes in patient's parents | at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephane BEZIEAU, PU-PH, Principal Investigator — Nantes University Hospital